CLINICAL TRIAL: NCT03724669
Title: A Multi-center Real-world Study of Benzodiazepines and Z-drugs Prescription in Psychiatric Clinic, and the Effectiveness of Electronic Interventions on Their Standardized Prescription of These Drugs
Brief Title: A Study of the Effectiveness of Electronic Interventions on the Standardized Prescription Benzodiazepines and Z-drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Second Xiangya Hospital of Central South University (Other); West China Hospital (Other); Suzhou Psychiatric Hospital, The Affiliated Guangji Hospital of Soochow University (Unknown); Wuhan Mental Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NZhong-001
Record Dates: First submitted 2018-10-28; First posted 2018-10-30 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2020-06

CONDITIONS: Bcenzodiazepines, Abuse, Retrospective Study, Focus Groups, Real-world Study
MeSH Terms: interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- waiting list (Placebo Comparator)
  Interventions: Behavioral: waiting list
- Benzodiazepines and Z-drugs knowledge (Experimental)
  Interventions: Behavioral: benzodiazepines related knowledge intervention

INTERVENTIONS:
Behavioral: waiting list — After the study ends, they will have access to receive the educational texts and view the online lectures.
  Arms: waiting list
Behavioral: benzodiazepines related knowledge intervention — participants receiving 11 articles pushing and 3 online lectures through the electronic interventions App, once a week, last for 3 months
  Arms: Benzodiazepines and Z-drugs knowledge

SUMMARY:
A retrospective surveys and group interviews focusing on the prescription and abuse of benzodiazepines will be carried out in China. Based the results of retrospective surveys and group interviews and guidelines of benzodiazepines and Z-drugs standardized use, a real-world randomized control trial of would be carried to evaluate the effectiveness of the intervention of using electronic content push in reducing the use rate of psychiatric BZDs and Z-drugs and improving clinical efficiency.

DETAILED DESCRIPTION:
Benzodiazepines (BZDs) and Z-drugs are commonly used sedative and hypnotic drugs in psychiatry. A small number of studies have suggestted that there may be improper use or even abuse in recent years. Long-term use of BZDs and Z-drugs may have the risk of impairing memory, respiratory depression, and increasing accidents risk. At present, there is no risk investigation on psychiatric BZDs and Z-drugs abuse in China, and many psychiatric practitioners lack of knowledge on the standard use of BZDs and Z-drugs. The aim of this study was to understand the use of benzodiazepines in psychiatric outpatient clinics in China and to develop a BZDs and Z-drugs standardized use electronic intervention guidebook and to verify the effectiveness of this electronic intervention in reducing the use of BZDs and Z-drugs in psychiatric outpatient clinics and improving clinical efficiency. Through retrospective surveys and focus interview groups, the study was conducted to understand the use of BZDs and Z-drugs and related factors of abuse in psychiatric outpatient clinics in Shanghai, Hunan, Sichuan, Wuhan and Jiangsu provinces. Based on the consensus and guidelines of domestic experts, BZDs and Z-drugs standardized electronic intervention was used. The real-world randomized controlled research method was combined with electronic content push and periodic electronic evaluation to evaluate the effectiveness of the intervention in reducing the use rate of psychiatric BZDs and Z-drugs and improving clinical efficiency. The research can deeply understand the use of BZDs and Z-drugs in domestic psychiatry and form an effective BZDs and Z-drugs standardized electronic intervention manual, which will provide practical value for regulating domestic BZDs and Z-drugs in the future.

ELIGIBILITY:
Inclusion Criteria:

1. at least 3-year working experience as a psychiatrist;
2. provide outpatient services for at least 1 year with the frequency of more than once a week;
3. willingness to receive standardized electronic interventions on BZDs and Z-drugs prescription.

Exclusion Criteria:

1. will retire within six months;
2. refuse to extract their prescription information from the outpatient database.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
proportion of inappropriate BZDs and Z-drugs prescription | 3 months before and after the intervention
  The BZDs and Z-drugs prescription information of each psychiatrist within the baseline period (3 months before the intervention) and intervention period (0-3 month) will be extracted from the outpatient prescription database in each hospital. The inappropriate prescription is defined as overdose use (>40mg), long-term use (>90 days) or over-indications use.

SECONDARY OUTCOMES:
BZDs and Z-drugs related knowledge | baseline, 3 months, 6 months
  22-item self-made questionnaite about BZDs and Z-drugs related knowledge
Attitude towards BZDs and Z-drugs prescription | baseline, 3 months, 6 months
  14-item self-made questionnaite about attitude towards BZDs and Z-drugs prescription
Common adverse effects in prescribing patients | baseline, 3 months, 6 months
  8-item self-made questionnaite about common adverse effects in prescribing patients
Self-efficacy | baseline, 3 months, 6 months
  An adapted 10-item version of General Self-Efficacy Scale (GSES) will be used to measure participants' self-efficacy.
Utility of the electronic intervention | 3 month
  an online 17-item questionnaire to evaluate the intervention and utilization data will be automatically collected through the platform

CONTACTS AND LOCATIONS:
Overall Officials: Na Zhong, Doctor, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
The prescription data will not be shared with the public. However, if the intervention is effective, the educational materials will be released to the public.

REFERENCES:
- [Derived] Xu X, Ye Y, Wang X, Xu J, Li C, Wang G, Zhu Y, Jiang H, Zhong N. Effectiveness and utility of an electronic intervention for appropriate benzodiazepine and Z-drugs prescription in psychiatric clinics: protocol for a multicentric, real-world randomised controlled trial in China. BMJ Open. 2022 Apr 5;12(4):e055341. doi: 10.1136/bmjopen-2021-055341. PMID 35383066